CLINICAL TRIAL: NCT00622609
Title: A Single-blind, Single Dose, Placebo Controlled, First Time in Human Study to Assess the Safety, Tolerability and Pharmacokinetics of Ascending Doses of GSK249320 in Healthy Volunteers
Brief Title: Anti-MAG First Administration to Human
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAG103114
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Cerebrovascular Accident
Keywords: first time in human,; MAG; monoclonal antibody,; healthy subjects,; GSK249320,
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects receiving GSK249320A (Experimental): Eligible subjects will receive escalating doses of GSK249320A in cohort 1 to 6 with a starting dose of 0.04 milligrams/kilograms up to the maximum dose of 25 milligrams/kilograms, administered as a slow intravenous infusion over 1 hour on Day 1.
  Interventions: Drug: GSK249320A
- Subjects receiving placebo (Placebo Comparator): Eligible subjects will receive single dose of sodium chloride in cohort 1 to 6, administered as a slow intravenous infusion over 1 hour on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK249320A — GSK249320A intravenous infusion will be formulated as 100 milligrams/milliliters in 2 milliliters vials (filled to 1 milliliter), in phosphate buffer and delivered by a syringe and programmable pump.
  Arms: Subjects receiving GSK249320A
Drug: Placebo — Sodium chloride intravenous infusion will be given as matching placebo.
  Arms: Subjects receiving placebo

SUMMARY:
GSK249320 is a monoclonal antibody directed against myelin associated glycoprotein (MAG), a protein that inhibits axonal regeneration. GSK249320 acts as a MAG antagonist, and through this activity it is hypothesised that it will enhance recovery from neuronal degeneration following acute axonal injury, which occurs in spinal cord injury or stroke.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men or women of non-child bearing potential (i.e. post-menopausal or surgically sterile e.g. hysterectomy or bilateral oophorectomy). If necessary, postmenopausal status will be confirmed by serum FSH and oestradiol concentrations at screening. Surgical sterility will be defined as females who have had a documented hysterectomy or bilateral oophorectomy.
* Between 18 and 60 years of age inclusive.
* Body weight >/ 60 kg and BMI within the range 19-29.9 kg/m2 inclusive.
* Healthy as judged by responsible physician with no clinically significant abnormality identified on the medical or laboratory evaluation. A subject with a clinical abnormality or laboratory parameters outside the reference range for this age group may be included only if the Investigator considers that the finding will not introduce additional risk factors and will not interfere with the study procedures.
* A 12-lead ECG at pre-study screening which in the opinion of the Investigator or his/her designee has no abnormalities that will compromise safety in this study.
* Normal clinical neurological exam, normal QST results, and normal pattern of conduction latencies in medial, ulnar, sural, tibial and peroneal nerves at screening.
* Signed and dated written informed consent prior to admission to the study.
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.

Exclusion Criteria:

* Positive drug/ alcohol screen at screening or baseline.
* Positive pre-study HIV, Hepatitis B surface antigen or positive Hepatitis C antibody result at screening.
* History of acute neuronal injury (central or peripheral) within the previous 12 months, peripheral neuropathy or neuritis, neurodegenerative disorders or other neurological diseases, including conditions which are known or hypothesised to be associated with disruption in the blood-brain barrier (BBB).
* Considered to be at a high risk of developing a stroke including a history of carotid artery disease or surgery, transient ischaemic attacks, reversible ischaemic neurological deficits or other abnormalities of the brain vessels, including but not limited to berry aneurysms or arteriovenous malformations.
* History of regular alcohol consumption averaging >7 drinks/week for women or >14 drinks/week for men. One drink is equivalent to (12 g alcohol) = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of 80 proof distilled spirits) within 6 months of screening.
* Subjects who smoke 10 or more cigarettes per day. Subjects who smoke <10 cigarettes per day may be admitted into the study but will be asked to refrain from smoking for at least 24 hours before the planned day of admission into the unit. They will NOT be allowed to smoke during their stay in the unit.
* The subject is unable to abstain from strenuous physical activity for 72 h prior to each clinic visit where safety lab tests are conducted.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* Where participation in study would result in donation of blood in excess of 500 mL within a 56 day period.
* Previous exposure to humanised antibody therapy for any reason.
* Unwillingness of the male subjects to abstain from sexual intercourse with pregnant or lactating women from the time of the first dose of study medication until five half lives following administration of the dose of study medication. This may be increased depending on PK analysis during the study.
* Unwillingness of the male subject to use a condom/spermicide in addition to having their female partner use another form of contraception such as an intra-uterine device (IUD), diaphragm with spermicide, oral contraceptives, injectable progesterone, subdermal implants or a tubal ligation if the woman could become pregnant from the time of the first dose of study medication until five half lives following administration of the last dose of study medication. The duration of the period during which contraception must be practiced may be modified during the study, depending on data emerging from PK analysis. The mean half-life predicted for GSK249320 is 30 days
* Female subjects with positive urine/serum pregnancy test result at screening or prior to first dose
* Status as a "vulnerable" subject, defined by the US Food and Drug Administration (FDA) Code of Federal Regulations; 45 CFR, Section 46, Subparts B and C.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2007-08-01 (Actual); Primary Completion 2009-04-09 (Actual); Study Completion 2009-04-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of GSK249320 including: adverse events,vital signs,ECG,continuous lead II ECG monitoring,safety laboratory assessments,clinical assessment of peripheral nerve function,nerve conduction testing | Throughout study

SECONDARY OUTCOMES:
Pharmacokinetic parametersAnti-GSK249320 antibody titres | At various timepoints from pre-dose to Week 52 follow-up
Pharmacokinetic parameters of ascending single IV doses of GSK249320: Cinf, AUC(0-24), AUC(0-t) and AUC(0-inf) | At various timepoints from pre-dose to Week 52 follow-up
Anti-GSK249320 Antibody titres: serum samples will be collected for anti-drug (anti-GSK249320) antibody confirmation, titration and neutralization testing | At various timepoints from pre-dose to Week 52 follow-up
Non-compartmental pharmacokinetic parameters of GSK249320 : Tinf , lz, T1/2, CL and Vss | At various timepoints from pre-dose to Week 52 follow-up
Novel candidate biomarkers and subsequently discovered biomarkers of the biological response associated with the action of GSK249320 may be identified by application of: | At various timepoints from pre-dose to Week 52 follow-up
RNA transcriptome analysis of blood samples | At various timepoints from pre-dose to Week 52 follow-up
Proteome analysis of plasma samples | At various timepoints from pre-dose to Week 52 follow-up

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Baltimore, Maryland, United States
- GSK Investigational Site, Randwick, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Abila B, Cunningham E, Simeoni M. First-time-in-human study with GSK249320, a myelin-associated glycoprotein inhibitor, in healthy volunteers. Clin Pharmacol Ther. 2013 Feb;93(2):163-9. doi: 10.1038/clpt.2012.227. Epub 2012 Nov 16. PMID 23267856
- See also: Results for study MAG103114 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/MAG103114?search=study&study_ids=103114#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: MAG103114 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: MAG103114 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: MAG103114 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: MAG103114 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: MAG103114 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: MAG103114 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register